CLINICAL TRIAL: NCT00262964
Title: Obesity and Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: DK37948; R01DK037948 (NIH)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2010-06-28 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: non-alcoholic fatty liver disease; obesity; fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Niacin; Fenofibrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NAFLD-Niacin (Experimental): Subjects, having previously diagnosed with NAFLD, were given Niacin for 16 weeks. The dosage was 500mg/day for week 1, 1000mg/day for week 2, 1500mg/day for week three and 2000mg/day for weeks 4 through 16.
  Interventions: Drug: Niacin
- Control (No Intervention): Subjects were found to have intrahepatic triglyceride levels below the threshold for Non-Alcoholic Fatty Liver Disease (NAFLD). For this study that threshold was set at 10% intrahepatic triglyceride content as determined by magnetic resonance spectroscopy. These control subjects did not participate in any intervention. Only baseline features were characterized for this arm.
- NAFLD-fenofibrate (Experimental): Subjects diagnosed with NAFLD were randomized to fenofibrate, an oral medication, nightly for eight weeks. Subjects will be given a dose of 200mg/day.
  Interventions: Drug: fenofibrate
- NAFLD-placebo (Placebo Comparator): These subjects were diagnosed with Non-Alcoholic Fatty Liver Disease (NAFLD) and received an 8 week course of a placebo pill. Their baseline characteristics were averaged into the overall NAFLD baseline characteristics along with the baseline data for the two intervention groups.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Niacin — Subjects randomized to Niacin therapy will be treated with Niacin at night for 16 wks to reduce plasma free fatty acid concentrations. The dose of medication will be gradually increased: 500 mg/day during week 1, 1000 mg/day during week 2, 1500 mg/day during week 3, and 2000mg/day during weeks 4-16.
  Other Names: niaspan
  Arms: NAFLD-Niacin
Drug: fenofibrate — Subjects randomized to fenofibrate will be treated with 200 mgs per day for eight weeks.
  Other Names: Tricor
  Arms: NAFLD-fenofibrate
Drug: placebo — Subjects randomized to placebo will be treated with one placebo pill per day for eight weeks.
  Arms: NAFLD-placebo

SUMMARY:
The primary goal of this study is to provide a better understanding of: 1) the pathogenesis and pathophysiology of non-alcoholic fatty liver disease (NAFLD) in obese subjects, and 2) the effect of marked weight loss on the histologic and metabolic abnormalities associated with NAFLD. The following hypotheses will be tested:

1. obesity causes hepatic fat accumulation because of excessive fatty acid release from fat tissue and increased free fatty acid availability,
2. increased hepatic (liver) fat content causes insulin-resistant glucose (sugar) production by the liver and altered liver protein synthesis,
3. increased hepatic fat content causes increased lipid (fat) peroxidation, hepatic inflammation, necrosis and fibrosis, and
4. marked weight loss improves NAFLD once patients are weight stable.

DETAILED DESCRIPTION:
Obesity is a major risk factor for non-alcoholic fatty liver disease (NAFLD), which represents a spectrum of liver diseases. NAFLD is a major health problem in the US because of its high prevalence and causal relationship with serious liver abnormalities. However, the mechanism(s)responsible for developing NAFLD in obese persons and the effects on liver function are not known. This gap in knowledge has made it difficult to identify effective therapy. The results from these studies will lay the groundwork for the development of novel therapeutic interventions for NAFLD in obese patients.

ELIGIBILITY:
Inclusion Criteria:

All

* 18 - 45 years old
* Class I obesity, i.e. Body Mass Index (BMI) between 30 and 45.
* weight less than 300 lbs.

Exclusion Criteria:

* Active or previous infection with hepatitis B or C, as well as other liver disease.
* History of alcohol abuse
* Diabetes
* Medications that cause liver damage or steatosis.
* Women who are pregnant or lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2004-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Beginning and ending recruitment dates: Beginning - 10/20/04; Ending - 09/24/07. Recruitment occurred only at Washington University in St. Louis.
Pre-assignment Details: We screened 138 subjects. 80 would-be participants failed the screening. This was often due to not having Non-alcoholic Fatty Liver Disease. Other subjects were excluded due to use of various medications or the presence of some excluded disease such as type 2 diabetes. Of the 58 that passed screening 51 chose to enroll in the study.
Groups:
- NAFLD - Niacin: subjects diagnosed with NAFLD were randomized to a sixteen week regimen of niacin.
- NAFLD - Fenofibrate: Subjects diagnosed with NAFLD were randomized to an eight week regimen of fenofibrate
- Controls: Subjects with normal intrahepatic fat triglyceride(IHTG) levels (<10%). IHTG was measured using magnetic resonance spectroscopy and defined as the extrapolated ratio of triglyceride signal to water signal at time t = 0.
- NAFLD - no Drug: Subjects with elevated intrahepatic triglyceride (IHTG) levels (>10%) who were measured only once (baseline). These subjects did not undergo drug therapy, in contrast to the NAFLD-niacin and NAFLD-fenofibrate group subjects. IHTG was measured using magnetic resonance spectroscopy and defined as the extrapolated ratio of triglyceride signal to water signal at time t = 0.
Period: Overall Study
Arm/Group | NAFLD - Niacin | NAFLD - Fenofibrate | Controls | NAFLD - no Drug
Started | 11 | 11 | 17 | 12
Completed | 11 | 11 | 17 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Controls: Subjects with normal intra-hepatic triglyceride content (defined by less than 10% lipid to water signal in magnetic resonance spectroscopy).
- NAFLD: Subjects diagnosed with Non-Alcoholic Fatty Liver Disease(NAFLD). Determination of NAFLD was by magnetic resonance spectroscopy of intra-hepatic triglyceride content (defined by greater than 10% lipid to water signal). This group included subjects later randomized into the NAFLD-Niacin, NAFLD-Fenofibrate, and NAFLD-no intervention arms.
- Total: Total of all reporting groups
Arm/Group | Controls | NAFLD | Total
Number analyzed (Participants) | 17 | 34 | 51
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 34 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (3) | 45 (3) | 42 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 24 | 37
  Male | 4 | 10 | 14
Region of Enrollment [Number; unit: participants]
  United States | 17 | 34 | 51
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 35.11 (4.33) | 36.73 (4.66) | 36.19 (4.57)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 99.8 (11.6) | 104.1 (15.6) | 102.7 (14.4)
fat as percentage of total body composition [Mean (Standard Deviation); unit: percentage of total body weight] — fat as percentage of total body composition as characterized using whole body Dual Energy X-ray Absorptiometry (DEXA).
  percentage of total body weight | 42.1 (6.9) | 39.3 (6.0) | 40.3 (6.4)
plasma glucose level [Mean (Standard Deviation); unit: mg/dl] — fasting plasma glucose level
  mg/dl | 94.2 (6.0) | 96.0 (8.6) | 95.4 (7.8)
plasma insulin level [Mean (Standard Deviation); unit: mU/L] — fasting plasma insulin
  mU/L | 11.4 (4.5) | 21.2 (9.9) | 17.9 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Insulin Sensitivity Index (HISI)
Description: Hepatic insulin sensitivity, assessed as a function of glucose production rate and plasma insulin concentration. The Hepatic Insulin Sensitivity Index(HISI) is the reciprocal of glucose rate of appearance [10000/(μmol/min)] multiplied by insulin concentration[mU/L]. The 10000 in the formula is a conventional adjustment so that insulin sensitivity measures are more readable. As yet there is no normal range for HISI, since is a surrogate marker for hepatic insulin sensitivity that has not yet been validated.
Time Frame: baseline cross-sectional data
Population: number of subjects determined by power calculations. Analysis was per protocol. Intrahepatic triglyceride was determined by magnetic resonance spectroscopy.
Measure: Mean (Standard Error); unit: [10000/(μmol/min)x(mU/L)]
Groups:
- NAFLD: subjects with intra-hepatic triglyceride content greater than 10%.
- Controls: subjects with normal intra-hepatic triglyceride levels
Arm/Group | NAFLD | Controls
Number analyzed (Participants) | 34 | 17
[10000/(μmol/min)x(mU/L)] | 0.8 (0.14) | 1.4 (0.26)
Statistical Analysis 1: Comparison: NAFLD vs Controls; null hypothesis was no difference in hepatic insulin sensitivity between normal and high IHTG subjects; Test type: Superiority or Other; p < 0.019, t-test, 2 sided

2. Secondary Outcome: Very Low Density Lipoprotein - Triglyceride Production Rate
Description: Very low density lipoprotein triglyceride (VLDL-TG) production rate, a measure of hepatic secretion of VLDL-triglyceride per liter of plasma per minute (μmol/L/min).
Time Frame: baseline cross-sectional data
Measure: Mean (Standard Error); unit: μmol/L/min
Groups:
- NAFLD: Subjects with intrahepatic triglyceride content greater than 10% per Magnetic Resonance Spectroscopy
- Controls: subjects with normal levels of intra-hepatic trigleceride
Arm/Group | NAFLD | Controls
Number analyzed (Participants) | 34 | 17
μmol/L/min | 6.7 (0.5) | 3.8 (0.3)
Statistical Analysis 1: Comparison: NAFLD vs Controls; null hypothesis was that VLDL-TG production would not differ between the two groups; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — a priori threshold for significance was P<0.05

3. Primary Outcome: Percent Increase in Skeletal Muscle Insulin Sensitivity During Insulin Infusion.
Description: A precise measure of the ability of insulin to stimulate glucose uptake by skeletal muscle. Skeletal muscle insulin sensitivity, measured as the increase from baseline in skeletal muscle glucose uptake during insulin infusion(percentage)as part of a nine hour euglycemic hyperinsulinemic clamp study.
Time Frame: baseline cross-sectional data pre and post nine hour euglycemic clamp
Measure: Mean (Standard Error); unit: percent increase
Groups:
- NAFLD: Subjects with intrahepatic triglyceride signal greater than 10% per MR spectroscopy
Arm/Group | NAFLD | Controls
Number analyzed (Participants) | 34 | 17
percent increase | 173 (13) | 303 (23)
Statistical Analysis 1: Comparison: NAFLD vs Controls; null hypothesis was no difference in skeletal muscle insulin sensitivity between groups; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — a priori threshold for significance was set at p = 0.05

4. Primary Outcome: Adipose Tissue Insulin Sensitivity
Description: The ability of insulin to suppress the release of fatty acids from adipose tissue: Adipose tissue insulin sensitivity, measured as the suppression from baseline of free fatty acid release from adipose tissue (lipolysis) during insulin infusion as part of a nine hour euglycemic hyperinsulinemic clamp study.
Time Frame: baseline cross-sectional data pre and post nine hour euglycemic clamp
Measure: Mean (Standard Error); unit: percent decrease
Groups:
- NAFLD: Subjects with elevated intrahepatic triglyceride (>10% signal compared to H2O) measured by MR Spectroscopy.
- Controls: subjects with normal intrahepatic triglyceride levels
Arm/Group | NAFLD | Controls
Number analyzed (Participants) | 34 | 17
percent decrease | 66 (2) | 75 (1)
Statistical Analysis 1: Comparison: NAFLD vs Controls; null hypothesis was that there would be no difference in adipose tissue insulin sensitivity due to IHTG levels; Test type: Superiority or Other; p < 0.002, t-test, 2 sided

5. Primary Outcome: Hepatic Fat Content for Fenofibrate and Niacin Groups
Description: Hepatic fat content as measured by magnetic resonance spectroscopy. A PRESS sequence was used. The results from three 10 cubic centimeter voxels positioned within the liver were averaged. The measure is a ratio of triglyceride signal to total signal.
Time Frame: baseline to post intervention: 8 weeks (fenofibrate), 16 weeks (niacin)
Population: 10 (or more) subjects in each group would be sufficient for detecting changes in IHTG.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- NAFLD - Niacin: subjects given niacin for 16 weeks
Arm/Group | NAFLD - Fenofibrate | NAFLD - Niacin
Number analyzed (Participants) | 11 | 11
ratio
  Baseline | 23.2 (10.2) | 21.0 (10.4)
  8 wk (fenofibrate), 16 wk (niacin) | 23.6 (11.2) | 19.7 (8.9)
Statistical Analysis 1: Comparison: NAFLD - Fenofibrate; Student's t-test for paired samples was used to evaluate any difference between the two groups. The null hypothesis was that the IHTG percentage would be the same before and after treatment for subjects receiving fenofibrate; Test type: Superiority or Other; p = .301, t-test, 2 sided — A P-value < 0.05 was considered statistically significant; Treatment effects determined by repeated-measures ANOVA. When significant interactions between time and group were found, a Student's t-test was used
Statistical Analysis 2: Comparison: NAFLD - Niacin; A Student's t-test for paired samples was used to evaluate the effect of treatment. The null hypothesis was that the IHTG percentage for the NAFLD-niacin group at baseline and post-treatment would not change; Test type: Superiority or Other; p = .315, t-test, 2 sided — A P-value < 0.05 was considered statistically significant; [statistical method as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Very Low Density Lipoprotein Apolipoprotein B Production Rate
Description: VLDL-apolipoprotein B (apoB) concentrations were measured as part of a VLDL metabolism study utilizing stable isotope tracers. VLDL apoB production rate, a measure of hepatic secretion of VLDL-apolipoproteinB-100 per liter of plasma per minute.
Time Frame: baseline to post intervention: 8 weeks (fenofibrate), 16 weeks (niacin)
Measure: Mean (Standard Error); unit: nmol/l/min
Arm/Group | NAFLD - Fenofibrate | NAFLD - Niacin
Number analyzed (Participants) | 11 | 11
nmol/l/min
  Baseline | 0.5 (0.05) | 0.4 (0.04)
  8 wk (fenofibrate), 16 wk (niacin) | 0.4 (0.05) | 0.4 (0.11)
Statistical Analysis 1: Comparison: NAFLD - Niacin; a Student's t-test for paired samples was used to evaluate the effect of treatment. Null hypothesis was that VLDL-apoB would be the same before and after 16 weeks on niacin in subjects with NAFLD; Test type: Superiority or Other; p = 0.708, t-test, 2 sided — A P-value < 0.05 was considered statistically significant
Statistical Analysis 2: Comparison: NAFLD - Fenofibrate; A Student's t-test for paired samples was used to evaluate the effect of treatment. Null hypothesis was that VLDL-apoB would be the same before and after 8 weeks on fenofibrate in subjects with NAFLD; Test type: Superiority or Other; p = .022, t-test, 2 sided — A P-value < 0.05 was considered statistically significant

7. Secondary Outcome: Change From Baseline in VLDL-Tg Clearance Rate
Description: Very low density lipoprotein triglyceride (VLDL-Tg) clearance rate, a measure of VLDL-triglyceride removal from plasma per minute.
Time Frame: baseline to end of treatment: 8 weeks (fenofibrate), 16 weeks (niacin)
Measure: Mean (Standard Error); unit: (ml/min)
Groups:
- NAFLD - Fenofibrate: Subjects with intrahepatic triglyceride signal greater than 10% per MR spectroscopy given an eight week course of fenofibrate
- NAFLD - Niacin: subjects with elevated levels of intra-hepatic trigleceride given a 16 week course of niacin
Arm/Group | NAFLD - Fenofibrate | NAFLD - Niacin
Number analyzed (Participants) | 11 | 11
(ml/min)
  Baseline | 35 (9) | 34 (8)
  8 weeks (fenofibrate) or 16 weeks (niacin) | 56 (12) | 52 (23)
Statistical Analysis 1: Comparison: NAFLD - Fenofibrate; the null hypothesis was that fenofibrate would not change the VLDL-Tg clearance rate; Test type: Superiority or Other; p = .020, t-test, 2 sided
Statistical Analysis 2: Comparison: NAFLD - Niacin; the null hypothesis was that niacin would not change the VLDL-Tg clearance rate; Test type: Superiority or Other; p = .358, t-test, 2 sided — a priori threshold for significance was <0.05

8. Secondary Outcome: Change From Baseline in VLDL-Tg Production Rate
Description: VLDL-TG production rate, a measure of hepatic secretion of VLDL-triglyceride per liter of plasma per minute.
Time Frame: baseline to end of treatment: 8 weeks (fenofibrate), 16 weeks (niacin)
Measure: Mean (Standard Error); unit: (μmol/L/min)
Groups:
- NAFLD - Fenofibrate: Subjects with intrahepatic triglyceride signal greater than 10% per MR spectroscopy receiving fenofibrate for eight weeks.
- NAFLD - Niacin: subjects with elevated levels of intra-hepatic trigleceride (>10% signal by MR spectroscopy) given a 16 week course of niacin
Arm/Group | NAFLD - Fenofibrate | NAFLD - Niacin
Number analyzed (Participants) | 11 | 11
(μmol/L/min)
  Baseline | 6.4 (0.7) | 7.7 (1.6)
  8 weeks (fenofibrate) or 16 weeks (niacin) | 6.0 (0.6) | 4.5 (0.8)
Statistical Analysis 1: Comparison: NAFLD - Fenofibrate; Null hypothesis is that fenofibrate would not effect VLDL-Tg production rates; Test type: Superiority or Other; p = 0.758, t-test, 2 sided — a priori threshold for statistical significance was set at <0.05
Statistical Analysis 2: Comparison: NAFLD - Niacin; Null hypothesis is that niacin would not effect VLDL-Tg production rates; Test type: Superiority or Other; p = .023, t-test, 2 sided — the a priori threshold for statistical significance was set at <0.05

9. Secondary Outcome: Change From Baseline in Very Low-density Lipoprotein Triglyceride Concentration
Description: Change from baseline in very low-density lipoprotein triglyceride concentration (VLDL-Tg)
Time Frame: baseline to end of treatment: 8 weeks (fenofibrate), 16 weeks (niacin)
Measure: Mean (Standard Error); unit: mmol/l
Arm/Group | NAFLD - Fenofibrate | NAFLD - Niacin
Number analyzed (Participants) | 11 | 11
mmol/l
  Baseline | 1.09 (0.28) | 1.04 (0.24)
  8 weeks (fenofibrate) or 16 weeks (niacin) | 0.50 (0.10) | 0.64 (0.23)
Statistical Analysis 1: Comparison: NAFLD - Fenofibrate; Null hypothesis was that fenofibrate would not affect VLDL-Tg concentration. We compare the pre and post-treatment results of subjects receiving an 8 week course of fenofibrate; Test type: Superiority or Other; p = .024, t-test, 2 sided — the a priori threshold for statistical significance was p <0.05
Statistical Analysis 2: Comparison: NAFLD - Niacin; The null hypothesis was that niacin would not affect VLDL-Tg concentration. We compare the pre and post-treatment results of subjects receiving a 16 week course of niacin; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — the a priori threshold for statistical significance was p<0.05

10. Primary Outcome: Adipose Tissue Insulin Sensitivity in Fenofibrate and Niacin Groups
Description: The baseline and post-treatment measures of adipose tissue insulin sensitivity (ATIS) were compared. ATIS at both timepoints is the suppression from fasting levels of free fatty acid release from adipose tissue (lipolysis) during an insulin infusion as part of a euglycemic clamp study. It is the percent decrease from time zero to the end of the nine hour euglycemic hyperinsulinemic clamp
Time Frame: baseline to post intervention: 8 weeks (fenofibrate), 16 weeks (niacin)
Measure: Mean (Standard Error); unit: percent decrease
Arm/Group | NAFLD - Fenofibrate | NAFLD - Niacin
Number analyzed (Participants) | 11 | 11
percent decrease
  Baseline | 68 (4) | 63 (4)
  8 weeks (fenofibrate) or 16 weeks (niacin) | 69 (2) | 35 (10)
Statistical Analysis 1: Comparison: NAFLD - Fenofibrate; Null hypothesis was that fenofibrate would not affect adipose tissue insulin sensitivity. We compare the baseline and post-treatment results for adipose tissue insulin sensitivity in the subjects who received fenofibrate; Test type: Superiority or Other; p = .768, t-test, 2 sided — A priori threshold for significance was set for p<0.05
Statistical Analysis 2: Comparison: NAFLD - Niacin; Null hypothesis was that niacin would not affect adipose tissue insulin sensitivity. Here we compare the baseline and post-treatment adipose tissue insulin sensitivity results for subjects who received a 16 week course of niacin; Test type: Superiority or Other; p = .019, t-test, 2 sided — A priori threshold for significance was set for p<0.05

11. Primary Outcome: Change From Baseline in Skeletal Muscle Insulin Sensitivity
Description: Changes in skeletal muscle insulin sensitivity (SMIS). SMIS was measured as the increase in skeletal muscle glucose uptake from time zero to the end of a nine hour euglycemic clamp and insulin infusion study. This increase is the percentage change from time zero to end of insulin infusion at nine hours.
Time Frame: baseline to end of treatment: 8 weeks (fenofibrate), 16 weeks (niacin)
Measure: Mean (Standard Error); unit: percent increase
Arm/Group | NAFLD - Fenofibrate | NAFLD - Niacin
Number analyzed (Participants) | 11 | 11
percent increase
  Baseline | 188 (36) | 183 (22)
  8 weeks (fenofibrate) or 16 weeks (niacin) | 169 (28) | 142 (26)
Statistical Analysis 1: Comparison: NAFLD - Fenofibrate; The null hypothesis was that fenofibrate would not affect skeletal muscle insulin sensitivity. Here we compare the pre and post-treatment results in subjects receiving an 8 week course of fenofibrate; Test type: Superiority or Other; p = .318, t-test, 2 sided — The a priori threshold for significance was set at p<0.05
Statistical Analysis 2: Comparison: NAFLD - Niacin; The null hypothesis was that niacin would not affect skeletal muscle insulin sensitivity. Here we compare the pre and post-treatment results for subjects receiving a 16 week course of niacin; Test type: Superiority or Other; p = .025, t-test, 2 sided — The a priori threshold for significance was set at p<0.05

12. Primary Outcome: Change From Baseline in Hepatic Insulin Sensitivity Index
Description: Hepatic insulin sensitivity, assessed as a function of glucose production rate and plasma insulin concentration. The Hepatic Insulin Sensitivity Index (HISI) is measured as the reciprocal of glucose rate of appearance [10000/(μmol/min)] multiplied by insulin concentration[mU/L]. The 10000 in the formula is a conventional adjustment so that insulin sensitivity measures are more readable. As yet there is no normal range for HISI, since is a surrogate marker for hepatic insulin sensitivity that has not yet been validated.
Time Frame: baseline to end of treatment: 8 weeks (fenofibrate), 16 weeks (niacin)
Measure: Mean (Standard Error); unit: [10000/(μmol/min)x(mU/L)]
Groups:
- NAFLD - Fenofibrate: Subjects with elevated intrahepatic triglyceride given an eight week course of fenofibrate
Arm/Group | NAFLD - Fenofibrate | NAFLD - Niacin
Number analyzed (Participants) | 11 | 11
[10000/(μmol/min)x(mU/L)]
  Baseline | 0.7 (0.1) | 0.8 (0.4)
  8 weeks (fenofibrate) or 16 weeks (niacin) | 0.8 (0.1) | 0.5 (0.1)
Statistical Analysis 1: Comparison: NAFLD - Fenofibrate; The null hypothesis was that fenofibrate would not affect hepatic insulin sensitivity. Here we compare the pre and post-treatment results of subjects receiving an 8 week course of fenofibrate; Test type: Superiority or Other; p = .419, t-test, 2 sided — The a priori threshold for significance was set at p<0.05
Statistical Analysis 2: Comparison: NAFLD - Niacin; The null hypothesis was that niacin would not affect skeletal muscle insulin sensitivity. Here we compare the pre and post-treatment results of subjects receiving a 16 week course of niacin; Test type: Superiority or Other; p = .018, t-test, 2 sided — The a priori threshold for significance was set at p<0.05

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline testing through post-treatment testing. The "NAFLD - no drug" and control groups were only followed through the baseline testing.
Groups:
- NAFLD - Fenofibrate: Subjects diagnosed with NAFLD were randomized to an weight week regimen of fenofibrate
- NAFLD - Niacin: subjects with intra-hepatic triglyceride signal greater than 10% placed on daily niacin for 16 weeks. The dose of medication will be gradually increased according to the protocol of most clinical trials (59): 500 mg/day during wk 1, 1000 mg/day during wk 2, 1500 mg/day during wks 3, and 2000mg/day during wks 4-16.
- NAFLD - no Drug: subjects with elevated hepatic triglyceride who did not receive any drug intervention
- Controls: subjects with normal hepatic triglyceride.
Arm/Group | NAFLD - Fenofibrate | NAFLD - Niacin | NAFLD - no Drug | Controls
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 1/11 | 0/11 | 0/12 | 0/17
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAFLD - Fenofibrate (N=11) | NAFLD - Niacin (N=11) | NAFLD - no Drug (N=12) | Controls (N=17)
elevation of liver enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — assessment of liver dysfunction by ALT and/or AST counts in blood plasma

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No